CLINICAL TRIAL: NCT06476834
Title: A Phase IV, Open-label, Single-group, Single-dose Study Evaluating Deucravacitinib Concentrations in the Breast Milk and Plasma of Healthy Lactating Female Participants
Brief Title: A Study Evaluating Deucravacitinib Concentrations in the Breast Milk and Plasma of Healthy Lactating Female Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-1123
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Deucravacitinib Administration (Experimental)
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165; SOTYKTU®

SUMMARY:
The purpose of this study is to evaluate Deucravacitinib concentrations in the breast milk and plasma of healthy lactating female participants.

ELIGIBILITY:
Inclusion Criteria

* Healthy female participants without, in the opinion of the investigator, clinically significant deviation from normal in medical history, physical examination, ECGs, vital signs, and clinical laboratory determinations.
* Body mass index (BMI) of 18.0 kg/m2 to 35.0 kg/m2, inclusive, and body weight ≥ 50 kg (110 lb), at screening. Given participants are postpartum, BMI accommodation up to 35.0 kg/m2 may be expected.
* Has well-established lactation (ie, at least 4 weeks postpartum) and can produce stable milk product (ie, approximately 3 oz per 3 hours at screening) using the methods required for the study.
* Is willing to exclusively pump breast milk for the 72-hour post dose period of milk collection during CRU confinement, and not to breastfeed or provide milk to infant until after CRU discharge (72 hours post dose).

Exclusion Criteria

* Presence or history of any clinically relevant abnormality, condition, or disease (such as liver disease or abnormal liver function tests, or cardiovascular or pulmonary diseases) that, in the opinion of the investigator, may affect absorption, distribution, metabolism, or elimination of the study intervention, that would prevent the participant from participating in the study, or which places the participant at unacceptable risk if she were to participate in the study.
* Current or recent (within 3 months of study intervention administration) clinically significant gastrointestinal disease that, in the opinion of the investigator, could impact upon the absorption of study intervention.
* Presence or history of mastitis, breast surgery or trauma, or other breast conditions, which are considered clinically significant by the investigator and/or, in the investigator's opinion, may significantly impact breastfeeding or collection of milk from one or both breasts.
* History of biliary disorders, including Gilbert's syndrome or Dubin-Johnson disease, except for isolated gallbladder issues, which are not by themselves exclusionary.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants received study treatment at one site in the United States of America.
Pre-assignment Details: Total 8 participants received study medication.
Groups:
- Deucravacitinib 9 mg: Participants received Deucravacitinib at a dose of 9 mg once daily
Period: Overall Study
Arm/Group | Deucravacitinib 9 mg
Started (Started=Treated) | 8
Completed (Completed=Completing the Treatment Period) | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (6.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of BMS-986165 and BMT-153261 in Breast Milk
Description: Cmax is defined as the maximum observed concentration of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
ng/mL
  BMS-986165 | 211.0 (59.5)
  BMT-153261 | 74.09 (55.7)

2. Primary Outcome: Time of Maximum Observed Concentration (Tmax) of BMS-986165 and BMT-153261 in Breast Milk
Description: Tmax is defined as the time taken to reach the maximum observed concentration (Cmax) of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Median (Full Range); unit: Hour
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Hour
  BMS-986165 | 1.00 [1.00 to 3.00]
  BMT-153261 | 6.00 [3.00 to 6.00]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours [AUC(0-24)] of BMS-986165 and BMT-153261 in Breast Milk
Description: AUC(0-24) defined as the area under the concentration-time curve from time zero to 24 hours of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 up to 24 hours post dose
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
h*ng/mL
  BMS-986165 | 1656 (54.5)
  BMT-153261 | 1289 (58.7)

4. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of BMS-986165 and BMT-153261 in Breast Milk
Description: AUC(INF) defined as the area under the concentration-time curve from time zero extrapolated to infinite time of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
h*ng/mL
  BMS-986165 | 1876 (57.9)
  BMT-153261 | 1767 (61.6)

5. Primary Outcome: Average Concentration (Cavg) of BMS-986165 and BMT-153261 in Breast Milk
Description: Cavg defined as the average concentration of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
ng/mL
  BMS-986165 | 78.18 (57.9)
  BMT-153261 | 73.61 (61.6)

6. Primary Outcome: Amount Recovered Within 24 Hours of Dosing [AR (24)] of BMS-986165 and BMT-153261 in Breast Milk
Description: AR (24) defined as the amount recovered within 24 hours of dosing of BMS-986165 and BMT-153261 in breast milk.
Time Frame: From first dose day 1 up to 24 hours post dose
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 6
mg
  BMS-986165 | 0.05021 (102.8)
  BMT-153261 | 0.03393 (107.1)

7. Primary Outcome: Total Amount Recovered (AR) of BMS-986165 and BMT-153261 in Breast Milk
Description: AR defined as the total amount recovered of BMS-986165 and BMT-153261 in breast milk.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 6
mg
  BMS-986165 | 0.05395 (106.0)
  BMT-153261 | 0.04230 (116.8)

8. Primary Outcome: Milk-plasma Ratio (M/P) of BMS-986165 and BMT-153261
Description: M/P defined as milk-plasma ratio of BMS-986165 and BMT-153261.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Ratio
  BMS-986165 | 3.241 (50.9)
  BMT-153261 | 15.76 (57.7)

9. Primary Outcome: Average Estimated Daily Infant Dose
Description: Average estimated daily infant dose represents the total amount of study medication that an infant is expected to consume each day average from day 1 to day 4, based on available data.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/kg/day
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
mg/kg/day | 0.01586 (58.8)

10. Primary Outcome: Average Relative Infant Dose
Description: Average relative infant dose shows the estimated percentage of the mother's weight-adjusted dose of study medication that the infant consumes through breast milk over a 24-hour period. This was averaged from day 1 to day 4 based on available data.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Percentage | 12.11 (53.6)

11. Secondary Outcome: Maximum Observed Concentration (Cmax) of BMS-986165 and BMT-153261 in Plasma
Description: Cmax is defined as the maximum observed concentration of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
ng/mL
  BMS-986165 | 62.56 (24.5)
  BMT-153261 | 4.797 (36.9)

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of BMS-986165 and BMT-153261 in Plasma
Description: AUC(INF) defined as the area under the concentration-time curve from time zero extrapolated to infinite time of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
h*ng/mL
  BMS-986165 | 587.2 (26.6)
  BMT-153261: number analyzed (Participants) | 7
  BMT-153261 | 128.3 (36.6)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours [AUC(0-24)] of BMS-986165 and BMT-153261 in Plasma
Description: AUC(0-24) defined as the area under the plasma concentration-time curve from time zero to 24 hours of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 up to 24 hours post dose
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
h*ng/mL
  BMS-986165 | 511.0 (24.4)
  BMT-153261 | 81.79 (39.6)

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-T)] of BMS-986165 and BMT-153261 in Plasma
Description: AUC(0-T) defined as the area under the plasma concentration-time curve from time zero to time of last quantifiable concentration of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
h*ng/mL
  BMS-986165 | 575.1 (26.9)
  BMT-153261 | 104.5 (52.4)

15. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of BMS-986165 and BMT-153261 in Plasma
Description: Tmax is defined as the time taken to reach the maximum observed plasma concentration (Cmax) of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Median (Full Range); unit: Hour
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Hour
  BMS-986165 | 2.00 [2.00 to 2.00]
  BMT-153261 | 6.00 [6.00 to 10.0]

16. Secondary Outcome: Average Concentration (Cavg) of BMS-986165 and BMT-153261 in Plasma
Description: Cavg defined as the average plasma concentration of BMS-986165 and BMT-153261 in plasma.
Time Frame: First dose day 1 to day 4 up to 72 hours
Population: All Pharmacokinetic (PK) participants who have at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
ng/mL
  BMS-986165 | 24.47 (26.6)
  BMT-153261: number analyzed (Participants) | 7
  BMT-153261 | 5.346 (36.6)

17. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent Adverse event (TEAE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: From the dose of study medication through 30 days (assessed for up to 30 days)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Participants | 0

18. Secondary Outcome: Number of Participants With Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Blood samples were collected to assess the abnormalities in laboratory parameters.
Time Frame: From the dose of study medication through 30 days (assessed for up to 30 days)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Participants | 0

19. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 17
Time Frame: From the dose of study medication through 30 days (assessed for up to 30 days)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Participants | 0

20. Secondary Outcome: Number of Participants With Abnormal Physical Examinations Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 17
Time Frame: From the dose of study medication through 30 days (assessed for up to 30 days)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Participants | 0

21. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 17
Time Frame: From the dose of study medication through 30 days (assessed for up to 30 days)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Deucravacitinib 9 mg
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality, SAEs and Other AEs from the dose of study medication through 30 days (assessed for up to 30 days).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Deucravacitinib 9 mg
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT06476834/Prot_SAP_000.pdf